CLINICAL TRIAL: NCT04119011
Title: A Novel Approach to Manipulate Intestinal Homeostasis in Primary Dysmenorrhoea Women: a Randomised Controlled Trial
Brief Title: Probiotics in Women With Primary Dysmenorrhoea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: B-Crobes Marketing(M) Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Prof Dr Nur Azurah Abd Ghani, Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2018-204
Record Dates: First submitted 2019-09-30; First posted 2019-10-08 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Primary Dysmenorrhea
Keywords: probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: placebo and probiotic are labelled A or B, this is prepared by the manufacturer and blinded from the participant and investigator, the unblinding takes place only after completion of the data collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotic in powder form containing lactobacillus and bifidobacterium strains, sugar, milk powder and flavoring, taken 2 sachets daily for 3 months
  Interventions: Biological: Probiotic
- Placebo (Placebo Comparator): Placebo in powder form containing sugar, milk powder, flavoring, taken 2 sachets daily for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Probiotic — (Lactobacillus acidophilus, lactobacillus casei, lactobacillus lactis) and Bifidobacterium (Bifidobacterium bifidum, bifidobacterium longum, bifidobacterium infantis) lactose, sugar, milk powder, oligosaccharides, ascorbic acid, citric acid, maltodextrin, and orange flavor
  Arms: Probiotic
Other: Placebo — lactose, sugar, milk powder, oligosaccharides, ascorbic acid, citric acid, maltodextrin, and orange flavor
  Arms: Placebo

SUMMARY:
This study compares the effect of probiotics versus placebo in women with primary dysmenorrhoea

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing probiotics against placebo in women with primary dysmenorrhoea

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles between 21 to 45 days
* primary dysmenorrhoea only
* willing to consume sachets twice daily for 3 months

Exclusion Criteria:

* current Intrauterine Copper Device (IUCD) user
* recent hormonal (estrogen or progesterone) therapy in last 3 months
* on treatment for allergy such as antihistamine
* diarrhoea with dairy product
* often take drugs which may affect the test results (such as medicines treating constipation or digestive medicine such as laxatives or enema)
* any malignant tumor regardless of type or site

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
pain score before treatment (visual analog scale VAS) | baseline
  mean Visual Analog Score on scale 0 to 10, on day 2 of menses at baseline
pain score after treatment (visual analog scale VAS) | after 3 months of treatment
  mean Visual Analog Score on scale 0 to 10, on day 2 of menses after 3 months of treatment with probiotic/placebo
severity score before treatment (verbal rating score) | baseline
  mean Verbal Rating Score on scale 0 to 3, on day 2 of menses at baseline
severity score after treatment (verbal rating score) | after 3 months of treatment
  mean Verbal Rating Score on scale 0 to 3, on day 2 of menses after 3 months of treatment with placebo/probiotic
Quality of life before treatment (Physical and mental health score assessed by SF12v2 questionnaire) | baseline
  mean quality of life score using validated health survey questionnaire Short Form 12 version 2 (SF12v2) (permission obtained from primary author) Answers from each question will be calculated using formula into percentage of average physical health score and average mental health score, on scale 0 to 100 in which higher percentage represents higher quality of life, and score less than 50 represents poor quality of life
Quality of life after treatment (physical and mental health score assessed by SF12v2 questionnaire) | at 3 months after completed treatment with probiotic or placebo
  mean quality of life score using validated health survey questionnaire Short Form 12 version 2 (SF12v2) (permission obtained from primary author) Answers from each question will be calculated using formula into percentage of average physical health score and average mental health score, on scale 0 to 100 in which higher percentage represents higher quality of life, and score less than 50 represents poor quality of life
Frequency of Non-steroidal Anti-Inflammatory Drugs (NSAIDs) use between placebo and probiotic group | 3 months during treatment with probiotic or placebo
  mean number of Non-steroidal Anti-Inflammatory Drugs (NSAIDs) use per cycle

SECONDARY OUTCOMES:
Concentration of inflammatory markers pre-treatment | baseline
  mean concentration of serum pro-inflammatory markers on day 2 of menses (Interleukin-1,2,4,5,6,7,8,10,12p70,13,17, Tumour necrosis factor-alpha, Granulocyte Colony Stimulating Factor, and Regulated on activation normal T-cell expressed and secreted) all in pg/mL, reported individually in table form
Concentration of inflammatory markers post-treatment | At 3 months after commencement of treatment
  mean concentration of serum pro-inflammatory markers on day 2 of menses (Interleukin-1,2,4,5,6,7,8,10,12p70,13,17, Tumour necrosis factor-alpha, Granulocyte Colony Stimulating Factor, and Regulated on activation normal T-cell expressed and secreted) all in pg/mL, reported individually in table form
intestinal microbiota before and after treatment with probiotics | on date of randomization and at 3 month after completed treatment with probiotic or placebo
  Relative abundance of microbiome DNA in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nur Azurah Abd Ghani, Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
clinical data sheet containing demographics, data collection (pain score, quality of life questionnaire, pain diary)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 20 months

REFERENCES:
- [Derived] Zakaria IA, Mohammed Zain NA, Teik CK, Abu MA, Zainuddin AA, Abdul Aziz NH, Safian N, Mohd Mokhtar N, Raja Ali RA, Beng Kwang N, Mohamed Ismail NA, Hamizan MR, Ab Razak WS, Nur Azurah AG. The role of probiotics in improving menstrual health in women with primary dysmenorrhoea: A randomized, double-blind, placebo-controlled trial (the PERIOD study). Womens Health (Lond). 2024 Jan-Dec;20:17455057241234524. doi: 10.1177/17455057241234524. PMID 38444064